CLINICAL TRIAL: NCT03314987
Title: Nucleophilic Defense Against PM Toxicity
Brief Title: Nucleophilic Defense Against PM Toxicity (NEAT Trial)
Acronym: NEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Timothy Edward O'Toole, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20.0258; 5R01ES019217 (NIH)
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Air Pollution Toxicity
Keywords: air pollution; oxidative stress; intervention
MeSH Terms: interventions — Carnosine

STUDY DESIGN:
Intervention Model Description: placebo controlled, randomized, double-blind
Who Masked: Participant, Investigator
Masking Description: double blind (participant, investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Active Comparator): Each participant will be given a daily oral dose of 2 grams of carnosine for 12 weeks
  Interventions: Dietary Supplement: L-carnosine
- placebo group (Placebo Comparator): Each participant will be given a daily oral dose of 2 grams of placebo for 12 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: L-carnosine — a naturally occurring di-peptide
  Arms: intervention group
Other: placebo — an identically appearing supplement
  Arms: placebo group

SUMMARY:
Carnosine is a naturally occurring peptide found in high levels in skeletal muscle and the brain and is also available commercially as a dietary supplement. Since carnosine has anti-oxidant properties and air pollution exposure induces a state of oxidative stress, the purpose of this study is to see if those taking carnosine as a dietary supplement are protected from air pollution-induced oxidative stress and adverse cardiovascular outcomes.

DETAILED DESCRIPTION:
This is a placebo controlled, randomized, double-blind, interventional trial investigating the efficacy of carnosine in reducing the effects of particulate matter air pollution (PM2.5). A total of 240 participants from the Louisville metropolitan and neighboring areas will be randomized into two dietary supplement study groups - carnosine (n=120) versus placebo (n=120). Intervention of study dietary supplements will occur from May through September, when the levels of PM2.5.are highest in the Louisville, KY area. Study participants will be given a daily oral dose of total of 2 grams of carnosine (or placebo) for a total of 12 consecutive weeks (during May through September).

Urinary levels of carnosine will be used to screen and identify potential candidates with low carnosine levels. Those with levels less than the median levels of the population, will be invited to participate in the study. The following measurements will be performed - blood and urine sample collection, physical examination, arterial stiffness, physical function, and self-reported surveys on environmental exposure, sleep, diet, and exercise. Supplement intervention (carnosine or placebo) will be initiated at the time of Baseline Assessment and will continue for 12 weeks from that date. Two follow up visits will occur at 6 weeks and 12 weeks respectively after initiating supplementation.

This innovative clinical investigation will provide an insight into the pre and post intervention effects of a cheap, safe, and over-the-counter available dietary supplement in countering the effects of air pollution.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between 22-65 years of age of either gender and all ethnicities,
2. All genders and all ethnicities
3. Residing in or near the Louisville metropolitan area
4. Consumes some type of meat/fish at least once a month during the past 3 months
5. Carnosine levels below the median level of the population
6. Agrees to complete all study visits and follow study intervention regimen
7. Will be living in the study area throughout the study period, with no more than 1 week away from the study area.

Exclusion Criteria:

1. Consumed any dietary supplement more than 3 times per week in the past 4 weeks (one month)
2. Current / ongoing treatment for substance abuse
3. Currently undergoing treatment or have conditions which may cause participant to be immunosuppressed
4. Diseases Affecting Peripheral Cell Count (i.e. Autoimmune Diseases - Hashimoto, Rheumatoid Arthritis, SLE, Rheumatoid Arthritis, Sjogren syndrome, Ankylosing Spondylitis, Takayasu arteritis, Kawasaki disease, Polyarteritis nodosa.)
5. Diseases Affecting Bone Marrow capacity
6. Diagnosis of any active cancer
7. Recent organ / kidney transplant or replacement (Active/Long-Term Medications)
8. Type 1 Diabetes Mellitus
9. Untreated thyroid disease
10. Untreated anemia
11. Current acute infections (Influenza, fever, etc.)
12. HIV positive status
13. Active/current Hepatitis HepA, HepB or HepC or in past 6 months
14. Currently or planning to be Pregnant / lactating
15. Prisoners / vulnerable populations
16. Other medical conditions that compromise completion of study
17. Unwilling to provide consent

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E. O'Toole, Principal Investigator — University of Louisville
Locations (1):
- Clinical Trials Unit, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Toole TE, Hellmann J, Wheat L, Haberzettl P, Lee J, Conklin DJ, Bhatnagar A, Pope CA 3rd. Episodic exposure to fine particulate air pollution decreases circulating levels of endothelial progenitor cells. Circ Res. 2010 Jul 23;107(2):200-3. doi: 10.1161/CIRCRESAHA.110.222679. Epub 2010 Jul 1. PMID 20595651
- [Result] Barski OA, Xie Z, Baba SP, Sithu SD, Agarwal A, Cai J, Bhatnagar A, Srivastava S. Dietary carnosine prevents early atherosclerotic lesion formation in apolipoprotein E-null mice. Arterioscler Thromb Vasc Biol. 2013 Jun;33(6):1162-70. doi: 10.1161/ATVBAHA.112.300572. Epub 2013 Apr 4. PMID 23559625
- [Result] Pope CA 3rd, Bhatnagar A, McCracken JP, Abplanalp W, Conklin DJ, O'Toole T. Exposure to Fine Particulate Air Pollution Is Associated With Endothelial Injury and Systemic Inflammation. Circ Res. 2016 Nov 11;119(11):1204-1214. doi: 10.1161/CIRCRESAHA.116.309279. Epub 2016 Oct 25. PMID 27780829
- [Derived] Baba SP, Amraotkar AR, Hoetker D, Gao H, Gomes D, Zhao J, Wempe MF, Rice PJ, DeFilippis AP, Rai SN, Pope CA 3rd, Bhatnagar A, O'Toole TE. Evaluation of supplementary carnosine accumulation and distribution: an initial analysis of participants in the Nucleophilic Defense Against PM Toxicity (NEAT) clinical trial. Amino Acids. 2024 Aug 31;56(1):55. doi: 10.1007/s00726-024-03414-5. PMID 39215872
- [Derived] O'Toole TE, Amraotkar AA, DeFilippis AP, Rai SN, Keith RJ, Baba SP, Lorkiewicz P, Crandell CE, Pariser GL, Wingard CJ, Pope Iii CA, Bhatnagar A. Protocol to assess the efficacy of carnosine supplementation in mitigating the adverse cardiovascular responses to particulate matter (PM) exposure: the Nucleophilic Defense Against PM Toxicity (NEAT) trial. BMJ Open. 2020 Dec 28;10(12):e039118. doi: 10.1136/bmjopen-2020-039118. PMID 33372072

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only screened participants with the lowest levels of endogenous carnosine (n=299) were invited to participate in the full study.
Groups:
- L-carnosine: Each participant will be given a daily oral dose of 2 grams of carnosine for 12 weeks
  L-carnosine: a naturally occurring di-peptide
Period: Overall Study
Arm/Group | L-carnosine | Placebo Group
Started | 153 | 146
Completed | 140 (13 from this group did not complete the full study) | 133 (13 from this group did not complete the full study)
Not Completed | 13 | 13
Not completed — Lost to Follow-up | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- L-carnosine Group: Each participant will be given a daily oral dose of 2 grams of carnosine for 12 weeks
  L-carnosine: a naturally occurring di-peptide
- Total: Total of all reporting groups
Arm/Group | L-carnosine Group | Placebo Group | Total
Number analyzed (Participants) | 153 | 146 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 153 | 146 | 299
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.4) | 45.1 (12.4) | 44.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 84 | 173
  Male | 64 | 62 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 17 | 30
  White | 130 | 116 | 246
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 153 | 146 | 299
urinary carnosine levels [Mean (Standard Deviation); unit: nmol/mg creatinine] | 11.3 (26.6) | 12.7 (17.6) | 12.1 (22.1)

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Progenitor Cells
Description: circulating pro-angiogenic cells
Time Frame: 3 months
Population: For some participants in both groups, insufficient blood samples were collected or there were errors in processing and data collection. Thus, the n=130 for both groups does not match with number of participants in the study visit.
Measure: Mean (Standard Error); unit: # cells per CD41 minus cells
Arm/Group | L-carnosine | Placebo Group
Number analyzed (Participants) | 130 | 130
# cells per CD41 minus cells | 0.0025 (0.0004) | 0.0027 (0.0007)

2. Secondary Outcome: Augmentation Index
Description: index of arterial function
Time Frame: 3 months
Population: For some participants, this data could not be collected, so the n does not equal the total number of participants.
Measure: Mean (Standard Deviation); unit: percentage of pulse pressure
Arm/Group | L-carnosine Group | Placebo Group
Number analyzed (Participants) | 137 | 134
percentage of pulse pressure | 122.6 (10.8) | 121.4 (10.4)

3. Secondary Outcome: Endothelial Microparticles
Description: index of endothelial damage
Time Frame: Samples were collected from each participant at baseline, after ~6wk of intervention, and after ~12wk of intervention. Measurement will be performed on archived samples once assay is in place.
Measure: Mean (Standard Error); unit: microparticles per microliter
Groups:
- L-carnosine: Each participant will be given a daily oral dose of 2 grams of carnosine for 12 weeks
- Placebo: Each participant will be given a daily oral dose of 2 grams of placebo for 12 weeks
Arm/Group | L-carnosine | Placebo
Number analyzed (Participants) | 33 | 38
microparticles per microliter | 1057 (177) | 709 (69)

4. Secondary Outcome: Platelet Monocyte Aggregates
Description: percentage of CD14 events that are co-stained with CD41 (platelet glycoprotein GPIIb); also levels of CD62P (P-selectin) expression
Time Frame: 3 months
Population: For some participants, blood samples were not collected or there were errors in processing or data collection. Thus n=132 and 128 is less than total number of participants.
Measure: Mean (Standard Error); unit: percent of events
Arm/Group | L-carnosine | Placebo
Number analyzed (Participants) | 132 | 128
percent of events | 12.3 (0.65) | 10.8 (0.58)

ADVERSE EVENTS:
Time Frame: a total of 5 months, from initial screening until one month after study completion
Description: adverse events as per clinical trials definition
  Information on events collected from participant report and by clinical team
Arm/Group | L-carnosine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/146
Serious Adverse Events (participants affected / at risk) | 3/153 | 3/146
Other Adverse Events (participants affected / at risk) | 24/153 | 16/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L-carnosine Group (N=153) | Placebo Group (N=146)
diarhhea (Gastrointestinal disorders) | 1 | 0
yeast infection (Infections and infestations) | 1 | 0
anxiety/depression (Psychiatric disorders) | 0 | 1
hypotension (Cardiac disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-carnosine Group (N=153) | Placebo Group (N=146)
tingling sensation (Nervous system disorders) | 11 (11) | 3 (3)
nausea (Gastrointestinal disorders) | 13 (13) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT03314987/Prot_SAP_000.pdf